CLINICAL TRIAL: NCT02363504
Title: Focus on the Locus Coeruleus Network With 7 T MRI: Link to Memory (Dys)Function
Brief Title: The Locus Coeruleus and Memory
Acronym: LOCUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: NL51297.068.14
Record Dates: First submitted 2015-02-04; First posted 2015-02-16 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer's Disease
Keywords: Magnetic Resonance Imaging; Noradrenaline; locus coeruleus; memory
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Saliva samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy older controls: 7 Tesla MRI with memory task and non-invasive neurostimulation
  Interventions: Other: 7 Tesla MRI with memory task and non-invasive neurostimulation
- Prodromal Alzheimer's disease patients: 7 Tesla MRI with memory task and non-invasive neurostimulation
  Interventions: Other: 7 Tesla MRI with memory task and non-invasive neurostimulation

INTERVENTIONS:
Other: 7 Tesla MRI with memory task and non-invasive neurostimulation — This is not an intervention, we investigate the neural mechanisms

SUMMARY:
The cause of Alzheimer's disease, the most common form of dementia, remains unknown. Neuropathological studies suggest that a small area in the brainstem, the locus coeruleus, might be the site of the onset of the disease. This area is the sole source of noradrenalin to the brain, a neurotransmitter involved in arousal, but also cognitive functions. Animal and pharmacological studies have hinted towards an important role of this area in memory functioning. However, these studies were hampered by the limited spatial resolution, making it hard to clearly localize the locus coeruleus in the brain. New developments in brain imaging allow now to visualize the brain with stunning precision. Furthermore, a non-invasive new stimulation method, transcutaneous vagus nerve stimulation, is believed to excite the locus coeruleus and thereby influencing neuronal networks and memory functioning.

There are three aims in this project:

1. To investigate how the functional interaction between the locus coeruleus and other brain areas, in particular the medial temporal lobe areas, during memory processes (encoding, consolidation and retrieval) change with development of Alzheimer's disease.
2. To investigate associations between noradrenaline, memory performance and brain functioning. The investigators aim to investigate how acute noradrenalin levels change during the different memory processes and whether or not this is beneficial for performance. Furthermore, the investigators will investigate whether this interaction between noradrenalin, memory performance and brain functioning is different healthy older individuals (n =35) or patients with prodromal Alzheimer's disease (n =35).
3. To investigate the underlying neural network changes during transcutaneous vagus nerve stimulation. The investigators will focus on differences in functional connectivity between the locus coeruleus and the medial temporal lobe areas in healthy older individuals and prodromal Alzheimer's disease patients. An experimental condition will be compared with a sham condition in a pseudo-randomized cross-over design.

ELIGIBILITY:
Inclusion Criteria:

For the patients:

* diagnosis of prodromal Alzheimer's disease based on the latest research criteria (clinical assessment at the memory clinic : presence of at least a memory impairment, memory complaints expressed by the patient or informant, no problems in daily life functioning, no dementia and presence of biomarkers
* Clinical Dementia Rating score of 0.5 (
* Mini-Mental State Examination (MMSE) ≥ 23 and being mentally competent (in general, individuals with a MMSE ≥ 18 are considered mentally competent)
* Age: between 60 and 85 years old
* 50% female
* Right-handedness
* Average level of education
* Informed consent before participation in the study

For the healthy older individuals:

* Average neuropsychological test results, in accordance with normative data, corrected for age, education and gender
* No substantial memory complaints (according to the participant)
* Age: between 60 and 85 years old
* 50% female
* Right-handedness
* Average level of education
* Informed consent before participation in the study

Exclusion Criteria:

* Reduced vision
* Psychoactive medication use
* Abuse of alcohol and drugs
* Cognitive impairment due to alcohol/drug abuse or abuse of other substances
* Past or present psychiatric or neurological disorders (major depression, schizophrenia, bipolar disorder, psychotic disorder (or treatment for it), epilepsy, stroke, Parkinson's disease, multiple sclerosis, brain surgery, brain trauma, electroshock therapy, kidney dialysis, Menière's disease, brain infections)
* Major vascular disorders (e.g. stroke)
* Heart diseases or pacemakers
* Contraindications for scanning (e.g. brain surgery, cardiac pacemaker, metal implants, claustrophobia, body tattoos)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 35 healthy older individuals and 35 patients with prodromal Alzheimer's disease
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) response during a memory task | 60 minutes
  BOLD response contrasts during encoding and retrieval. For encoding: comparing neutral versus emotional, comparing old versus prodromal AD and the interaction emotional level by group. For retrieval: correctly remembered versus those incorrectly remembered; neutral versus emotional faces; lures, mistakes and hits. These contrasts will be investigated comparing both groups.
  BOLD responses during the memory task will also be compared across sessions (sham versus stimulation) for both groups.
  Consolidation: task-free, so the BOLD response in the locus coeruleus will be correlated with the BOLD response in any other voxel of the grey matter of the brain over time (seed-based resting-state analyses).
Performance on the memory task | 60 minutes
  Mean reaction times and accuracy levels during encoding and retrieval for emotional and neutral face-name associations and for old and prodromal AD patients.
  Mean reaction times and accuracy levels will also be compared across sessions: sham versus stimulation for both groups Mean reaction times and accuracy levels will also be correlated with BOLD responses during the memory task.
Noradrenalin levels during the memory task | 60 minutes
  Noradrenalin levels will be measured 7 times: double baseline, before encoding, after encoding, before retrieval, after retrieval and follow-up.
  Noradrenalin levels will be correlated with BOLD responses during the memory task.

SECONDARY OUTCOMES:
Grey matter volume of the locus coeruleus | 5 mintues
  manual measurement of the number of voxels of the locus coeruleus: to compare groups
shape properties of the locus coeruleus | 5 minutes
  Correspondence of the location between triangle meshes (shape of the locus coeruleus) will be compared between groups
Performance on neuropsychological tests | 30 minutes
  Total score on the mini-mental state examination, fluency test, letter-digit-substitution test, concept shifting task, stroop color word test and the word learning task will be compared across groups. For the stroop color word task and the concept shifting task we will also compare reaction times between both groups.
  These scores will be correlated to the grey matter volume of the locus coeruleus and the shape properties of the locus coeruleus.

OTHER OUTCOMES:
Basic descriptives | 15 minutes
  gender, date of birth, socio-economic status, educational level, medical history, medication use: will be used descriptively
Vascular measurements | 15 min
  Mean arterial blood pressure, cardiovascular risk factors and vascular pathology will be assessed descriptively and could also lead to exclusion of participants.
Alpha-peak frequency | 30 minutes
  the individual mean alpha-peak frequency will be assessed with rest EEG to determine stimulation parameters.
Side effects | 10 min
  via a questionnaire we will collect the level of side effects after stimulation (scale 1-5)
Blood pressure and heart rate | 20 minutes
  Blood pressure and heart rate will be measured before and after the sessions (seated and standing) in order to monitor response to the stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Frans Verhey, Prof, Study Director — Maastricht University Medical Centre
Locations (1):
- Maastricht University, Maastricht, Netherlands